CLINICAL TRIAL: NCT05947357
Title: Addressing LatinX Cancer Care Equity: Food for Health Equity
Brief Title: Food for Health Equity: Evaluation of a Nutrition Assistance Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 64256
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Food Insecurity; Food Assistance Quality Improvement Program; Latinx and minority patients
MeSH Terms: conditions — Neoplasms | interventions — Food Assistance

STUDY DESIGN:
Intervention Model Description: Patients as part of a nutrition assistance program will randomly receive food vouchers for $40.00 each month for use in the produce section of local grocery stores for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Assistance Program (Experimental): A total of 30 Latinx cancer patients on active cancer treatment who have screened positive for food insecurity will receive a $40.00 voucher for use each month for 6 months for nutrition assistance in the produce section of local grocery stores after enrollment in the program.
  Interventions: Other: Nutrition Assistance Program

INTERVENTIONS:
Other: Nutrition Assistance Program — Patients will receive in the intervention group a $40.00 per month voucher for 6 months for use in the produce section of a local grocery store.

SUMMARY:
This study seeks to evaluate whether a nutrition assistance quality improvement program for patients with cancer and food insecurity receiving active treatment at Pacific Cancer Care will have reductions in food insecurity.

DETAILED DESCRIPTION:
This study seeks to evaluate the effectiveness and patient satisfaction with a nutrition assistance quality improvement program in which a randomly selected 30 patients will receive a food voucher with $40.00 each month for 6 months for use in the produce section at local grocery stores in the county. The primary outcome is understanding whether this program is effective at reducing food insecurity among patients being treated for cancer and will provide key insights that may guide program expansion or improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient Participants must be undergoing or starting treatment for cancer at the Pacific Cancer Care clinic who screen positive for food insecurity using at 2-item screener, speak English or Spanish, have capacity to consent (e.g. no dementia or other cognitive impairment), are Latinx or another racial and ethnic minority group OR low income, have public insurance, OR are insured by an agricultural company sponsored health insurance

Exclusion Criteria:

* Patients will be ineligible if they do not have a current cancer diagnosis, cannot communicate in English or Spanish, are deemed ineligible to consent, are under 18 years of age, are not Latinx or another racial/ethnic minority OR are not low income OR are not publicly insured, uninsured, or do not have health insurance from an agricultural company

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Food Insecurity | Baseline to 6 months
  Assessed using the validated 2-item Hunger Vital Sign, administered to participants at time of enrollment and again at 6-months post-enrollment. Responses to questions "often" and "sometimes" versus "never" which are considered affirmative responses. One or more affirmative responses indicate food insecurity.

SECONDARY OUTCOMES:
Food Security | Baseline to 6 months
  Assessed using the validated United States Department of Agriculture (USDA) Six Item Food Security Survey will be administered to participants at time of enrollment and again at 6-months post-enrollment.
  Rabbit MP, Hales LJ, Reed-Jones M. Survey Tools. Accessed October 16, 2024, 2024. https://www.ers.usda.gov/topics/food-nutrition-assistance/food-security-in-the-u-s/survey-tools/#six
Health-related quality of life (HRQOL) | Baseline to 6 months
  Assessed using the 27-item validated Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire. The questionnaire has a scale of 0-108, with higher scores correlating with better quality of life.
  Cella DF, Tulsky DS, Gray G, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. Journal of clinical oncology : official journal of the American Society of Clinical Oncology. 1993/03// 1993;11(3):570-579. doi:10.1200/jco.1993.11.3.570
Financial Toxicity | Baseline to 6 months
  Assessed using the 12-item Comprehensive Score for Financial Toxicity - Functional Assessment of Chronic Illness Therapy (COST-FACIT) score. Scores range from 0-44 with higher scores correlating with better financial well-being.
  de Souza JA, Yap BJ, Wroblewski K, et al. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. Feb 1 2017;123(3):476-484. doi:10.1002/cncr.30369
Health-related social needs | Baseline to 6 months
  Assessed using the validated 13-item the Accountable Health Communities (AHC) Health-Related Social Needs Screening Tool from the Center for Medicare and Medicaid Services. Each question is scored from 1 to 5, based on the response option, scores are tallied. Totals range from 4 to 20. Higher scores indicate greater health-related social needs.
Satisfaction with the intervention | Baseline to 6 months
  Assessed using a 5-question tool where patients rated their satisfaction with the quality of intervention components and likelihood to recommend it to others. Scores were summed and higher scores indicated greater satisfaction.
Treatment Adherence | Baseline to 6 months
  Using a 1-item dichotomous question on treatment adherence. Adherence to cancer treatment was defined as having no missed scheduled clinic or treatment visits, which was abstracted from the electronic health record.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States